CLINICAL TRIAL: NCT06789965
Title: Randomized Clinical Trial Comparing Two Surgical Techniques for the Treatment of Type III Obesity (BMI 40-50 kg/m2): Single Anastomosis Duodeno-ileal Bypass With Sleeve Gastrectomy (SADI-S) and Roux-en-Y Gastric Bypass (RY-GBP)
Brief Title: Comparison of Two Surgical Techniques for Treatment of Type III Obesity (BMI 40-50 kg/m2): Single Anastomosis Duodenoileal Bypass With Sleeve Gastrectomy and Roux-en-Y Gastric Bypass.
Acronym: BYPSADIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HCB/2024/0752
Record Dates: First submitted 2024-12-16; First posted 2025-01-23 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Obesity
Keywords: obesity; sadi-s; ry-gbp; weight loss; metabolic complications; sadis; gbp; rygbp; bariatric surgery
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SADI-S (Experimental): The complete dissection of the antrum and the first portion of the duodenum is performed up to the limit of the gastroduodenal artery. The right gastric artery is dissected, clipped, and sectioned at its root. A vertical gastrectomy is created using a 38F Foucher tube with staplers. Next, the duodenum is sectioned with a stapler, and the resection of the greater gastric curvature is completed. Then, from the left side of the patient, 250 cm is measured from the ileocecal valve, where the duodenoileal anastomosis will be performed. This anastomosis is carried out with the surgeon positioned again between the patient's legs. A manual end-to-side anastomosis with two layers of monofilament is performed. Finally, the vertical gastrectomy and the duodenoileal anastomosis are verified using intraoperative endoscopy or a methylene blue and air test. The gastrectomy specimen is removed through the left pararectal trocar incision. A drain will only be placed in cases of special technical diff
  Interventions: Procedure: SADI-S
- RY-GBP (Active Comparator): In the case of RY-GBP, first, the lesser gastric curvature is dissected between the cardia and the angular incisura, accessing the gastric transcavity. A horizontal gastric transection is performed using the first firing of a stapler. A gastric reservoir is created through successive firings with a 38F Foucher tube stapler. Next, 100 cm of the biliopancreatic limb is measured, where the manual or semi-mechanical gastrojejunostomy will be performed, with an end-to-side anastomosis using a stapler and manual closure of the loop. Then, 150 cm of the alimentary limb is measured, and a side-to-side jejunojejunostomy is created. A section is made between the two anastomoses. The mesenteric opening and the Petersen space are closed with a continuous non-absorbable suture. The anastomosis is verified using intraoperative endoscopy or a methylene blue and air test. A drain will only be placed in cases of special technical difficulty or intraoperative complications.
  Interventions: Procedure: RY-GBP

INTERVENTIONS:
Procedure: SADI-S — In the case of SADI-S, the complete dissection of the antrum and the first portion of the duodenum is performed up to the limit of the gastroduodenal artery. The right gastric artery is dissected, clipped, and sectioned at its root. A vertical gastrectomy is created using a 38F Foucher tube with staplers. Next, the duodenum is sectioned with a stapler, and the resection of the greater gastric curvature is completed. Then, from the left side of the patient, 250 cm is measured from the ileocecal valve, where the duodenoileal anastomosis will be performed. This anastomosis is carried out with the surgeon positioned again between the patient's legs. A manual end-to-side anastomosis with two layers of monofilament is performed. Finally, the vertical gastrectomy and the duodenoileal anastomosis are verified using intraoperative endoscopy or a methylene blue and air test. The gastrectomy specimen is removed through the left pararectal trocar incision. A drain will only be placed in cases of s
  Arms: SADI-S
Procedure: RY-GBP — In the case of RY-GBP, first, the lesser gastric curvature is dissected between the cardia and the angular incisura, accessing the gastric transcavity. A horizontal gastric transection is performed using the first firing of a stapler. A gastric reservoir is created through successive firings with a 38F Foucher tube stapler. Next, 100 cm of the biliopancreatic limb is measured, where the manual or semi-mechanical gastrojejunostomy will be performed, with an end-to-side anastomosis using a stapler and manual closure of the loop. Then, 150 cm of the alimentary limb is measured, and a side-to-side jejunojejunostomy is created. A section is made between the two anastomoses. The mesenteric opening and the Petersen space are closed with a continuous non-absorbable suture. The anastomosis is verified using intraoperative endoscopy or a methylene blue and air test. A drain will only be placed in cases of special technical difficulty or intraoperative complications.
  Arms: RY-GBP

SUMMARY:
Roux-en-Y gastric bypass (RY-GBP) is one of the surgical techniques most widely used for the treatment of obesity. Long series of operated patients published in the literature have demonstrated its safety and efficacy. It consists on the reduction of the size of the stomach and joining it (anastomosis) with the small bowel to reduce the absorption of calories.

Single anastomosis duodenoileal with sleeve gastrectomy is an increasingly used surgical technique that is a simplification of the duodenal switch. It consists on the reduction of the stomach to a tube (sleeve gastrectomy) and an anastomosis between the duodenum and the small bowel. It has been demonstrated as a effective technique and it is supported by the international scientific societies.

There are no data that indicate a superiority of one technique over the other. The objective of this study is to analyze if there are differences between the two techniques in terms of postoperative weight control and gastroesophageal reflux at short, medium and long term.

DETAILED DESCRIPTION:
Obesity is being considered an epidemic of our century. It directly or indirectly contributes as the leading cause of non-traumatic death in the Western population and is progressively reaching developing countries as well. In Spain, recent epidemiological studies estimate that over 15% of the population is at least overweight, and nearly 5% has morbid obesity. The treatment of obesity is multidisciplinary, ranging from lifestyle and dietary changes to surgery. Among all available treatments, the only truly cost-effective option for patients with morbid obesity is bariatric surgery. The beneficial effects go far beyond weight loss, as it has been shown to reduce and improve comorbidities, enhance quality of life, lower cardiovascular risk, and even reduce mortality in individuals affected by obesity.

Duodenal switch (DS) has proven to be the most effective surgical procedure for treating morbid obesity and its comorbidities. However, it currently represents a small percentage of bariatric surgeries performed worldwide, likely due to its technical complexity and the risk of long-term complications. In an effort to simplify the DS technique, in 2007, Drs. Sánchez-Pernaute and Torres introduced the Single Anastomosis Duodeno-Ileal bypass with Sleeve gastrectomy (SADI-S). The omega reconstruction, which avoids the distal ileo-ileal anastomosis, aims to decrease surgical time and reduce postoperative risks. The SADI-S involves a vertical gastrectomy (VG) and a duodeno-ileal anastomosis with preservation of the pylorus, jejunal exclusion, and an original total common channel of 200 cm, standardized later to 250 or 300 cm to minimize the risk of nutritional deficiencies. The SADI-S can be performed as a primary direct surgery, planned in two stages, or as a revisional surgery in case of weight loss failure after VG. Various prospective studies presented on SADI-S show weight loss results and reduction of comorbidities similar to those of large historical series of DS.

The Roux-en-Y gastric bypass (RY-GBP) is currently considered the gold standard of bariatric surgery. It involves creating a small gastric reservoir and a Roux-en-Y gastrojejunostomy.

his is a well-standardized technique with large cohorts of patients followed over the long term, which has demonstrated safety and efficacy in weight control, resolution of metabolic comorbidities, as well as improvement in life expectancy and quality of life. Furthermore, it is the best technique for preventing or treating gastroesophageal reflux (GERD), due to its small gastric reservoir and rapid emptying. However, it has potential specific complications resulting from the non-preservation of the pylorus and mesenteric partitioning: anastomotic ulcer, early or late dumping syndrome, hypoglycemia, and abdominal pain associated with internal hernias. All of these complications are rare but much more frequent after an RY-GBP than after a SADI-S.

Currently, there is only one ongoing study comparing the efficacy and safety of SADI-S with RY-GBP. This is SADISLEEVE (ClinicalTrials.gov ID NCT03610256), a French multicenter randomized study that has several methodological limitations in its design: it includes both patients undergoing primary and revisional surgery, without BMI restrictions and with varying lengths of limbs.

The present prospective randomized study aims to compare SADI-S with RY-GBP. It includes patients with a BMI between 40 and 50 kg/m² for whom gastric bypass would be indicated at the participating centers. Patients who do not meet the requirements for bariatric surgery, as well as those with contraindications for hypoabsorptive or mixed surgery, are excluded.

The project has two objectives: a) efficacy: to compare the percentage of weight lost at 2 and 5 years after the two surgical procedures; b) safety: to assess the percentage of serious complications at 2 and 5 years. Routine follow-up controls from both Endocrinology and Dietetics, as well as General Surgery, will be used for both.

The most relevant secondary objective is to compare quality of life, for which SF-12 questionnaires will be systematically administered, along with the most likely factors affecting it: resolution of comorbidities, symptoms of GERD, abdominal pain, dumping syndrome, hypoglycemia, diarrhea, and need for supplementation. Gastroscopy and esophageal pH-impedance measurement will also be performed before the operation and at 2 and 5 years post-surgery.

Other secondary objectives include comparing short-term complications and studying nutritional and metabolic deficits of both procedures in the medium and long term. For the study of morbidity and mortality, the electronic medical records of the patients will be used, classifying immediate postoperative events (up to 30 days post-intervention) according to the Clavien-Dindo classification. The analysis of comorbidity evolution will involve monitoring factors related to metabolic risk in these patients before the intervention and annually thereafter, utilizing the infrastructure of the patient follow-up protocol. Finally, the analysis of metabolic and nutritional deficits will be conducted through comparative analysis of the annual analytical data systematically collected during the follow-up of the intervened patients.

Main Hypothesis: The Single Anastomosis Duodeno-Ileal bypass (SADI-S) is associated with greater efficacy (higher percentage of weight loss) and similar safety (equal or lower percentage of serious complications) at two and five years post-surgery compared to gastric bypass (RY-GBP) in patients with grade III morbid obesity (BMI between 40 and 50 kg/m²).

Secondary Hypotheses:

1. SADI-S is associated with lower incidence of digestive symptoms: dumping syndrome, hypoglycemia, and abdominal pain.
2. SADI-S is associated with better quality of life than RY-GBP.
3. RY-GBP is associated with a lower risk of GERD and a higher risk of anastomotic ulcer.
4. The complication rates of both techniques in the immediate postoperative period (up to 30 days post-intervention) are similar.
5. SADI-S achieves higher rates of resolution of metabolic syndrome comorbidities: type 2 diabetes mellitus (T2DM), hypertension (HT), dyslipidemia (DL), and sleep apnea (SA).
6. Patients undergoing SADI-S and RY-GBP require similar supplementation to compensate for nutritional deficits in the short, medium, and long term.
7. Baseline eating habits are related to weight loss at 2 and 5 years within each of the two patient groups.
8. Differences in acid and bile reflux occur between the two techniques, which can be objectively measured with functional tests such as pH-metry, impedance measurement, and bilitec.

ELIGIBILITY:
Inclusion Criteria:

* BMI 40 - 50 Kg/m2
* Candidates to mixed bariatric surgery

Exclusion Criteria:

* < 18 years.
* > 60 years.
* BMI < 40 Kg/m2
* BMI > 50 Kg/m2.
* Non-candidates to mixed bariatric surgery.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 450 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2030-08-01 (Estimated)

PRIMARY OUTCOMES:
% of patients with Total weight loss at 2 years > 30% | 2 years after intervention
  % of patients with Total weight loss at 2 years > 30%
% of patients with Total weight loss at 5 years > 30% | 5 years after intervention
  % of patients with Total weight loss at 5 years > 30%
Short term postoperative complications | From intervention to the end of the short term at 30 days after surgery.
  Complications classified as Clavien-Dindo III or IV (requiring reintervention, endoscopic or radioguided interventional treatment, or admission to the ICU).
Middle to long-term postoperative complications | From 30 days after intervention to the end of the study 5 years after the intervention.
  In the medium to long term, any complication that requires reintervention, endoscopic or radioguided interventional treatment, ICU admission, maintained parenteral or enteral nutrition, or specific parenteral treatment is included. This encompasses complications attributable to bariatric surgery, such as intestinal obstruction, internal hernia, diarrhea, hypoglycemia, dumping syndrome, malnutrition, ulcer, and GERD. Reintervention due to incisional hernia, cholecystectomy, or causes unrelated to bariatric surgery is excluded.

SECONDARY OUTCOMES:
Digestive symptoms at 2 years after surgery | From the intervention up to 2 years after surgery
  Prevalence of digestive symptoms (dumping syndrome, hypoglycemia, GERD, bowel habits, and abdominal pain) at 2 years measured using the following scales: ARTS for dumping syndrome, GERD Q for gastroesophageal reflux disease, Bristol and Wexner scales for bowel habits, QoL SF-12 for abdominal pain)
Digestive symptoms at 5 years after surgery | From the 2nd year until the end of the follow-up 5 years after the intervention.
  Prevalence of digestive symptoms (dumping syndrome, hypoglycemia, GERD, bowel habits, and abdominal pain) at 5 years measured using the following scales: ARTS for dumping syndrome, GERD Q for gastroesophageal reflux disease, Bristol and Wexner scales for bowel habits, QoL SF-12 for abdominal pain)
Endoscopic findings at 2 years | From the intervention up to 2 years after surgery
  Prevalence of endoscopic findings(esophagitis, ulcer, gastritis, bile lakes) at 2 years
Postoperative morbidity and mortality | From the intervention up to 90 days after surgery
  Postoperative morbidity and mortality (30 and 90 days after surgery)
Resolution of metabolic comorbidities at 2 years | From the intervention up to 2 years after surgery
  Resolution of metabolic comorbidities (T2DM, hypertension, dyslipidemia, and sleep apnea) at 2 years.
Resolution of metabolic comorbidities at 5 years | 5 years after intervention
  Resolution of metabolic comorbidities (T2DM, hypertension, dyslipidemia, and sleep apnea) at 5 years
Quality of life | From the intervention to the end of the study 5 years after the intervention.
  Difference on the total puntuation of the quality of life scales SF-12 at 2 and 5 years measured using the QoL scale SF-12.
Metabolic and nutritional deficits at 2 and 5 years | From the intervention to the end of the follow-up at 5 years after surgery.
  Prevalence of metabolic and nutritional deficits at 2 and 5 years measured using BARSCORE
Eating habits | Before the intervention up to 5 years after the intervention.
  Difference in the total count of the Dutch Behaviour Questionnaire of eating habits before the intervention, at 2 years and 5 years after surgery measured using the Dutch Behaviour Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Osorio, PhD, Principal Investigator — General & Digestive Surgery Department, ICMDM, Clinic Barcelona
Locations (1):
- Hospital Clinic Barcelona, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared upon request to the principal investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 1 year after publication with no end date.
Access Criteria: The requests for IPD sharing will be reviewed by the IP and a committee of the IPs from the different centers. Access will be granted for systematic reviews and metaanalysis.

REFERENCES:
- [Background] Arts J, Caenepeel P, Bisschops R, Dewulf D, Holvoet L, Piessevaux H, Bourgeois S, Sifrim D, Janssens J, Tack J. Efficacy of the long-acting repeatable formulation of the somatostatin analogue octreotide in postoperative dumping. Clin Gastroenterol Hepatol. 2009 Apr;7(4):432-7. doi: 10.1016/j.cgh.2008.11.025. Epub 2008 Dec 13. PMID 19264574
- [Background] Scarpellini E, Arts J, Karamanolis G, Laurenius A, Siquini W, Suzuki H, Ukleja A, Van Beek A, Vanuytsel T, Bor S, Ceppa E, Di Lorenzo C, Emous M, Hammer H, Hellstrom P, Laville M, Lundell L, Masclee A, Ritz P, Tack J. International consensus on the diagnosis and management of dumping syndrome. Nat Rev Endocrinol. 2020 Aug;16(8):448-466. doi: 10.1038/s41574-020-0357-5. Epub 2020 May 26. PMID 32457534
- [Background] Clapp B, Hahn J, Dodoo C, Guerra A, de la Rosa E, Tyroch A. Evaluation of the rate of marginal ulcer formation after bariatric surgery using the MBSAQIP database. Surg Endosc. 2019 Jun;33(6):1890-1897. doi: 10.1007/s00464-018-6468-6. Epub 2018 Sep 24. PMID 30251139
- [Background] Nandipati KC, Bremer KC. Bariatric Surgery Emergencies in Acute Care Surgery. Surg Clin North Am. 2023 Dec;103(6):1113-1131. doi: 10.1016/j.suc.2023.05.013. Epub 2023 Jul 1. PMID 37838459
- [Background] van Beek AP, Emous M, Laville M, Tack J. Dumping syndrome after esophageal, gastric or bariatric surgery: pathophysiology, diagnosis, and management. Obes Rev. 2017 Jan;18(1):68-85. doi: 10.1111/obr.12467. Epub 2016 Oct 17. PMID 27749997
- [Background] Pletch A, Lidor A. GERD after Bariatric Surgery: A Review of the Underlying Causes and Recommendations for Management. Curr Gastroenterol Rep. 2024 Apr;26(4):99-106. doi: 10.1007/s11894-024-00919-7. Epub 2024 Feb 14. PMID 38353898
- [Background] Olbers T, Beamish AJ, Gronowitz E, Flodmark CE, Dahlgren J, Bruze G, Ekbom K, Friberg P, Gothberg G, Jarvholm K, Karlsson J, Marild S, Neovius M, Peltonen M, Marcus C. Laparoscopic Roux-en-Y gastric bypass in adolescents with severe obesity (AMOS): a prospective, 5-year, Swedish nationwide study. Lancet Diabetes Endocrinol. 2017 Mar;5(3):174-183. doi: 10.1016/S2213-8587(16)30424-7. Epub 2017 Jan 6. PMID 28065734
- [Background] Syn NL, Cummings DE, Wang LZ, Lin DJ, Zhao JJ, Loh M, Koh ZJ, Chew CA, Loo YE, Tai BC, Kim G, So JB, Kaplan LM, Dixon JB, Shabbir A. Association of metabolic-bariatric surgery with long-term survival in adults with and without diabetes: a one-stage meta-analysis of matched cohort and prospective controlled studies with 174 772 participants. Lancet. 2021 May 15;397(10287):1830-1841. doi: 10.1016/S0140-6736(21)00591-2. Epub 2021 May 6. PMID 33965067
- [Background] Gronroos S, Helmio M, Juuti A, Tiusanen R, Hurme S, Loyttyniemi E, Ovaska J, Leivonen M, Peromaa-Haavisto P, Maklin S, Sintonen H, Sammalkorpi H, Nuutila P, Salminen P. Effect of Laparoscopic Sleeve Gastrectomy vs Roux-en-Y Gastric Bypass on Weight Loss and Quality of Life at 7 Years in Patients With Morbid Obesity: The SLEEVEPASS Randomized Clinical Trial. JAMA Surg. 2021 Feb 1;156(2):137-146. doi: 10.1001/jamasurg.2020.5666. PMID 33295955
- [Background] Angrisani L, Santonicola A, Iovino P, Ramos A, Shikora S, Kow L. Bariatric Surgery Survey 2018: Similarities and Disparities Among the 5 IFSO Chapters. Obes Surg. 2021 May;31(5):1937-1948. doi: 10.1007/s11695-020-05207-7. Epub 2021 Jan 12. PMID 33432483
- [Background] Salminen P, Gronroos S, Helmio M, Hurme S, Juuti A, Juusela R, Peromaa-Haavisto P, Leivonen M, Nuutila P, Ovaska J. Effect of Laparoscopic Sleeve Gastrectomy vs Roux-en-Y Gastric Bypass on Weight Loss, Comorbidities, and Reflux at 10 Years in Adult Patients With Obesity: The SLEEVEPASS Randomized Clinical Trial. JAMA Surg. 2022 Aug 1;157(8):656-666. doi: 10.1001/jamasurg.2022.2229. PMID 35731535
- [Background] Lind RP, Ghanem M, Teixeira AF, Jawad MA, Osorio J, Lazzara C, Sobrino L, Ortiz-Ciruela D, de Gordejuela AGR. Single- Versus Double-Anastomosis Duodenal Switch: Outcomes Stratified by Preoperative BMI. Obes Surg. 2022 Dec;32(12):3869-3878. doi: 10.1007/s11695-022-06315-2. Epub 2022 Oct 24. PMID 36279044
- [Background] Osorio J, Lazzara C, Admella V, Franci-Leon S, Pujol-Gebelli J. Revisional Laparoscopic SADI-S vs. Duodenal Switch Following Failed Primary Sleeve Gastrectomy: a Single-Center Comparison of 101 Consecutive Cases. Obes Surg. 2021 Aug;31(8):3667-3674. doi: 10.1007/s11695-021-05469-9. Epub 2021 May 12. PMID 33982240
- [Background] Finno P, Osorio J, Garcia-Ruiz-de-Gordejuela A, Casajoana A, Sorribas M, Admella V, Serrano M, Marchesini JB, Ramos AC, Pujol-Gebelli J. Single Versus Double-Anastomosis Duodenal Switch: Single-Site Comparative Cohort Study in 440 Consecutive Patients. Obes Surg. 2020 Sep;30(9):3309-3316. doi: 10.1007/s11695-020-04566-5. PMID 32240495
- [Background] Hess DS, Hess DW. Biliopancreatic diversion with a duodenal switch. Obes Surg. 1998 Jun;8(3):267-82. doi: 10.1381/096089298765554476. PMID 9678194
- [Background] Hess DS, Hess DW, Oakley RS. The biliopancreatic diversion with the duodenal switch: results beyond 10 years. Obes Surg. 2005 Mar;15(3):408-16. doi: 10.1381/0960892053576695. PMID 15826478
- [Background] Hess DS; 2004 ABS Consensus Conference. Biliopancreatic diversion with duodenal switch. Surg Obes Relat Dis. 2005 May-Jun;1(3):329-33. doi: 10.1016/j.soard.2005.03.217. No abstract available. PMID 16925243
- [Background] Gagner M, Matteotti R. Laparoscopic biliopancreatic diversion with duodenal switch. Surg Clin North Am. 2005 Feb;85(1):141-9, x-xi. doi: 10.1016/j.suc.2004.10.003. PMID 15619535
- [Background] Feng JJ, Gagner M. Laparoscopic biliopancreatic diversion with duodenal switch. Semin Laparosc Surg. 2002 Jun;9(2):125-9. PMID 12152155
- [Background] Biron S, Hould FS, Lebel S, Marceau S, Lescelleur O, Simard S, Marceau P. Twenty years of biliopancreatic diversion: what is the goal of the surgery? Obes Surg. 2004 Feb;14(2):160-4. doi: 10.1381/096089204322857492. PMID 15018742
- [Background] Biertho L, Lebel S, Marceau S, Hould FS, Lescelleur O, Moustarah F, Simard S, Biron S, Marceau P. Perioperative complications in a consecutive series of 1000 duodenal switches. Surg Obes Relat Dis. 2013 Jan-Feb;9(1):63-8. doi: 10.1016/j.soard.2011.10.021. Epub 2011 Nov 15. PMID 22189411
- [Background] Batista Marchesini J. A Safer and Simpler Technique for the Duodenal Switch : To the Editor: Obes Surg. 2007 Aug;17(8):1136. doi: 10.1007/s11695-007-9192-1. No abstract available. PMID 17973180
- [Background] Baltasar A, Bou R, Miro J, Bengochea M, Serra C, Perez N. Laparoscopic biliopancreatic diversion with duodenal switch: technique and initial experience. Obes Surg. 2002 Apr;12(2):245-8. doi: 10.1381/096089202762552430. PMID 11975221
- [Derived] Osorio J, Lazzara C, Guimaraes M, Torres A, Turrado-Rodriguez V, Ibarzabal A, Sobrino L, Nora M, Vilarrassa N, de Hollanda A, Rubio-Herrera MA, Vidal J, Moize V, Yarnoz C, Fernandez-Falop I, Portillo M, Sanchez-Pernaute A. A randomized open-label multicentre clinical trial comparing single-anastomosis duodenal switch (SADI-S) versus Roux-en-Y gastric bypass for the treatment of severe obesity: BYPSADIS study protocol. Scand J Surg. 2025 Oct 17:14574969251385873. doi: 10.1177/14574969251385873. Online ahead of print. PMID 41104829